CLINICAL TRIAL: NCT00318097
Title: Histamine Responsiveness in Patients With McCune-Albright Syndrome
Brief Title: Histamine Responsiveness in McCune-Albright Syndrome
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: KBR (Unknown)
Other Study IDs: 03 11-116
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: McCune-Albright Syndrome
Keywords: McCune Albright Syndrome; Histamine regulation
MeSH Terms: conditions — Fibrous Dysplasia, Polyostotic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- MAS patients: patient with clinical diagnosis of MAS
- controls: age matched, tanner stage matched controls

SUMMARY:
McCune-Albright syndrome (MAS) is a syndrome caused by a genetic mutation that causes a specific protein in the body called a G protein to be constantly active. Children with McCune-Albright syndrome classically have early puberty, areas of increased skin pigmentation, and bone lesions resulting from the constant activity of the specific protein involved.

Histamines are known to play a role in allergies and related allergic problems. The effects of histamines are controlled by the same G protein that is overly active in McCune-Albright syndrome. Thus, one could predict that patients with McCune-Albright may be at high risk for allergic problems. To date, no studies have documented any form of histamine excess or allergic difficulties in patients with McCune-Albright syndrome. However, the investigators have made the observation that a high percentage of their patients with MAS exhibit a range of allergic symptoms, from mild symptoms, to severe, life-threatening symptoms.

The purpose of this study is to demonstrate increased histamine response by using a histamine skin test in patients with MAS. If increased reactions to histamines can be documented in MAS patients when compared to controls, severe and potentially life threatening allergic reactions in children with MAS could be anticipated and avoided.

DETAILED DESCRIPTION:
Objectives of this study are to determine if:

1. Patients with McCune-Albright syndrome differ from unaffected controls in wheal and flare response to histamine and codeine.
2. Affected skin will differ from unaffected skin in wheal and flare response to histamine and codeine.
3. IgE and IL-4 levels in MAS patients differ from normal controls.

Specific Aims:

1. Compare the skin response of MAS patients to normal controls using standard histamine and codeine skin testing.
2. Compare skin testing response in MAS patients with known standards for skin testing. Compare response to histamine and codeine skin testing in MAS patient's affected (café-au-lait) skin to unaffected (normal) skin.
3. Compare IgE and IL-4 levels in patients with MAS to controls.

Background:

The McCune-Albright syndrome (MAS) is a genetic disorder characterized by constitutive activation of the Gαs proteins involved in the adenylyl cyclase enzyme. The disease is now known to be caused by a genetic mutation, commonly a substitution of histadine or cysteine for arginine at amino acid 201 in the Gαs protein. Adenylyl cyclase, with its formation of cyclic AMP (cAMP), works as a second messenger for many cellular and hormonal events. Clinically, MAS is characterized classically by precocious puberty, café-au-lait skin markings, and bone lesions termed polyostotic fibrous dysplasia. Other conditions that represent overactivity of receptor-coupled adenylate cyclase include hyperthyroidism resulting from activation of the TSH receptor, hypercortisolism (CRH and ACTH receptor activation), acromegaly (GHRH receptor activation), among others. Clinical heterozygosity of affected individuals is explained by mosaicism of the mutation.

The H2 histamine receptor is also coupled to the Gαs protein. Release of histamine from mast cells is primarily responsible for immediate hypersensitivity reaction in the skin. Clinical observations of our patients with MAS suggest increased responsiveness to histamine. We speculate that this results from upregulation of Gαs coupled to H2 receptor. In our identified patients, this has been manifested as asthma, chronic hives, dermatographism, contact hypersensitivities, drug reactions, ulcers, as well as anaphylactic reactions to seafood, dyes, and latex. Approximately 75% of our patients with MAS exhibit one or more of the aforementioned reactions. Anaphylaxis has occurred in three separate patients.

Interleukin-4 (IL-4) is also released from immune cells in response to histamine. This cytokine response is mediated by H2 receptor activation and activation of Gαs. IL-4 is required for function and production of IgE, another important mediator of hypersensitivity reactions. Two of our MAS patients with allergy symptoms have additionally demonstrated markedly elevated IgE levels.

Codeine is a very effective agent in causing release of histamine from mast cells and is commonly used in addition to histamine. We plan to use codeine as well as histamine skin testing to evaluate histamine response. Comparison of codeine responses between the MAS patients and unaffected controls will be made. Age and sex do not exert major effects on histamine responsiveness. Only infants and adults over the age of 50 have been noted to have decreased responsiveness in comparison to other age groups. Menstrual cycles in females have been noted to cause slight variation with increased dermal reactivity around ovulation and lower reactivity during the menses. Because most girls with McCune-Albright have irregular menses it will be difficult to time skin testing with the menstrual cycle. Therefore, we will record the date of last menstrual period for each female patient and control.

Excessive histamine responsiveness has not been a reported association of the MAS complex. Even though data are available, MAS patients could be predicted to be at risk for vigorous histamine response, because histamine acts via Gαs.

Study Design:

This will be a single center controlled study of histamine response in children with MAS compared to unaffected subjects. No investigational drug/device/biologic agent will be employed.

Subject Selection Criteria:

1. Expected sample size: 10 McCune-Albright patients and 20 controls.
2. Patients will be recruited for the study during endocrinology clinic visits. Most patients with MAS are seen at least every 6 months. Families of patients with MAS tend to be medically sophisticated, as MAS can be a severe, chronic, multisystem disease. We estimate that at least 80% of our 13-14 known patients will consent to participate. A control group will also be recruited.
3. Inclusion criteria: Children with MAS ranging from toddlers to young adults. Diagnosis of MAS will be made on a clinical basis. Blood testing is not helpful in this condition, as bone marrow progenitor cells with the Gαs mutation display a survival disadvantage. All patients are mixed chimeras, as this mutation is lethal if it occurs in germline cells. Patients who exhibit two or more of the following clinical findings fit the diagnosis of MAS:

   1. GnRH independent precocious puberty
   2. Polyostotic fibrous dysplasia
   3. Café-au-lait spots with Coast of Maine borders and respect for the midline.
   4. Non-autoimmune hyperthyroidism. Ten controls will also be recruited from family members of patients with MAS with no known allergies. An additional control group of ten unrelated subjects, also with no known allergies, will be recruited from the Endocrine Clinic for comparison.
4. Exclusion criteria:

   1. Any MAS patient or control who has not or cannot discontinue any home regimens of antihistamines or glucocorticoids (including inhaled steroids) at least seven days prior to skin testing.
   2. Any MAS patient or control on tricyclic antidepressants within two weeks prior to skin testing.

Study Groups:

No specific treatment is being investigated in this study.

Observations/Measurements:

Patients will be asked to have discontinued any usual home regimens of antihistamines and/or glucocorticoids for seven days prior to skin testing. First each participant will undergo a single blood draw to obtain levels of IgE and IL-4. We will utilize commercially available ELISA kits for human IL-4. We have published extensively using ELISA methods. Quantitative IgE levels will be performed in our lab.

Children with MAS and controls will undergo standard pin-prick skin testing procedures with dilutions of histamine, codeine, and a saline control solution to assess skin wheal and flare response in order to objectively assess hypersensitivity and/or responsiveness. Skin testing specifically involves placing a drop of histamine solution on the skin surface. A needle is then penetrated gently into the epidermis. The same procedure will be used for codeine and saline. Tests will be spaced at least 2 cm apart to avoid false reactions. Testing will include two standard sites for skin testing, i.e. arm and back, for all participants. An area of skin with café-au-lait formation and its normal skin counterpart will be tested on the patients with MAS. The normal controls will undergo skin testing at a matched area. Testing will be performed in the Allergy Clinic by a trained allergy fellow or attending. Wheal and flare responses will be documented 20 minutes after the skin tests are administered. The wheal and flare response will be outlined in ink, and the image will be transferred to hypoallergenic transparent tape and placed on a data collection sheet for measurement. The longest and orthogonal erythema diameters are measured and summed. Sum of wheal diameters will be determined in a similar manner. Previous studies have shown that a standard wheal and flare response yields a sum of 7.0 cm ± 1.25 cm.

After testing is complete, participants will then be given a dose of antihistamine (Zyrtec) and topical calamine lotion to pin prick areas to decrease irritation. There will be careful monitoring for extreme hypersensitivity or anaphylaxis as is the usual standard of care when testing children for allergies. However, classic systemic allergic reactions are caused by protein allergens. As histamine and codeine are not protein compounds, a systemic allergic reaction would not be expected. An epinephrine pen will be on hand for use if such an unusual reaction occurs.

Significance:

Currently there is no literature stating that children with McCune-Albright syndrome display an increased responsiveness to histamine. If this study shows that MAS patients indeed do have increased histamine responsiveness, risk for severe allergic reactions could be anticipated. Life threatening events could be potentially averted by having MAS patients carry epinephrine pens and/or by treating these patients with antihistamines.

Power analysis:

A published report of standard wheal and flare responses to histamine demonstrates that the sum of the longest (A) and orthogonal (B) (determined by the midpoint of A, labeled X) [Σ =A+B] diameter of the wheal and flare response to histamine was 7.0 cm ± 1.25 cm. (mean ± S.D.) Assuming that McCune-Albright patients will display a mean wheal and flare response 50% greater in diameter compared to controls, and using an alpha level of 0.05; testing of 10 patients will provide an 84% power to detect differences between patients and controls.

ELIGIBILITY:
Inclusion Criteria:

* Children with MAS ranging from toddlers to young adults.
* Diagnosis of MAS will be made on a clinical basis. Blood testing is not helpful in this condition, as bone marrow progenitor cells with the Gαs mutation display a survival disadvantage. All patients are mixed chimeras, as this mutation is lethal if it occurs in germline cells.
* Patients who exhibit two or more of the following clinical findings fit the diagnosis of MAS:

  * GnRH independent precocious puberty
  * Polyostotic fibrous dysplasia
  * Café-au-lait spots with coast of Maine borders and respect for the midline.
  * Non-autoimmune hyperthyroidism.
* Ten controls will also be recruited from family members of patients with MAS with no known allergies. An additional control group of ten unrelated subjects, also with no known allergies, will be recruited from the Endocrine Clinic for comparison.

Exclusion Criteria:

* Any MAS patient or control who has not, or cannot, discontinue(d) any home regimens of antihistamines or glucocorticoids (including inhaled steroids) at least seven days prior to skin testing.
* Any MAS patient or control on tricyclic antidepressants within two weeks prior to skin testing.

Max Age: 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2007-08-01 (Actual); Study Completion 2007-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela L Turpin, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States